CLINICAL TRIAL: NCT06350565
Title: A Clinical Pharmacological Study of Dose Halving of Dexamethasone in Pregnant Women With Preterm Labour With Preterm Birth at Greater Than or Equal to 34 Gestational Weeks (34GW+)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhao Yangyu, Vice director of Drug Clinical Trial Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX20240104
Record Dates: First submitted 2024-03-13; First posted 2024-04-05 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Distress Syndrome of Newborn
Keywords: Dexamethasone; Pregnancy; Quantitative pharmacology
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Half-dose study (Other): A total of 24 Chinese pregnant subjects with 34+0-35+6 GW requiring dexamethasone treatment for preterm labour with preterm prematurity in China were planned to be enrolled in this study. A total of 12 subjects receiving 5 mg dexamethasone (intramuscular injection, q12h, 4 doses) were enrolled in the full-dose group; 12 subjects receiving 2.5 mg dexamethasone (intramuscular injection, q12h, 4 doses) were enrolled in the half-dose group.
  Interventions: Drug: Dexamethasone
- An exploratory study (Other): This study was planned to enrol 24 pregnant women with 34+0-38+6 GW preterm labour with confirmed gestational diabetes mellitus (GDM) or diabetes mellitus in combination with pregnancy in a dose exploratory study in this population. A total of 12 subjects were enrolled in the full-dose group to receive 5 mg dexamethasone (intramuscular injection, q12h, 4 doses) and 12 subjects were enrolled in the half-dose group to receive 2.5 mg dexamethasone (intramuscular injection, q12h, 4 doses).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — This clinical study will plan to enrol 24 Chinese pregnant subjects with 34+0-35+6GW preterm preterm labour requiring dexamethasone treatment and 24 pregnant women with 34+0-38+6GW preterm preterm labour and a diagnosis of gestational diabetes mellitus (GDM) or diabetes mellitus in combination with pregnancy, each of them randomly divided into 2 groups requiring 4 doses of dexamethasone intramuscularly (half-dose of 2.5 mg, normal dose of 5 mg) for two days as well as two active blood acquisitions. During the recruitment and screening phase, the purpose of the trial, the study protocol, and the trial procedure were described in detail so that the subjects were fully informed and participated voluntarily, and the compliance of the subjects in the conduct of the trial was improved.

SUMMARY:
This study plans to conduct a DEX dose halving study and a normal dose study in 34+0-35+6 GW women with preterm preterm labour. In addition, this study plans to conduct a DEX dose halving study and a normal dose study in 34-38+6 GW preterm pregnant women with GDM or diabetic co-pregnancy to explore the feasibility of dose halving in pregnant women with diabetes mellitus.

DETAILED DESCRIPTION:
Two studies will be conducted both of which are single-centre, open clinical studies. It is proposed to collect maternal blood, umbilical vein blood and placental tissue from pregnant women treated with dexamethasone, which excludes early placental detachment, use of surfactant, severe intrauterine haemorrhage, or pregnant women who meet the conditions of the exclusion criteria. Determination and implementation of dexamethasone treatment regimen will be carried out by clinicians in accordance with the treatment guidelines, and the collection of samples will be carried out in the form of opportunistic blood sampling or placenta collection after normal diagnostic and therapeutic operations of pregnant women except for 2 active collections of blood after dosing; this study will not interfere with the normal maternal pregnancy, labour and diagnostic and therapeutic processes.

Half-dose study: A total of 24 Chinese pregnant subjects with 34+0-35+6 GW requiring dexamethasone treatment for preterm labour with preterm prematurity in China were planned to be enrolled in this study. A total of 12 subjects receiving 5 mg dexamethasone (intramuscular injection, q12h, 4 doses) were enrolled in the full-dose group; 12 subjects receiving 2.5 mg dexamethasone (intramuscular injection, q12h, 4 doses) were enrolled in the half-dose group.

EXPLORATORY STUDY: This study was planned to enrol 24 pregnant women with 34+0-38+6 GW preterm labour with confirmed gestational diabetes mellitus (GDM) or diabetes mellitus in combination with pregnancy in a dose exploratory study in this population. A total of 12 subjects were enrolled in the full-dose group to receive 5 mg dexamethasone (intramuscular injection, q12h, 4 doses) and 12 subjects were enrolled in the half-dose group to receive 2.5 mg dexamethasone (intramuscular injection, q12h, 4 doses).

ELIGIBILITY:
Inclusion Criteria:

Common criteria for half-dose studies and exploratory studies:

1. Age 18-40 years (inclusive);
2. Body mass index (BMI) 18.5-27.9 kg/m2 (inclusive).
3. risk of preterm labour and use of dexamethasone for fetal lung maturation.

Half-dose study-specific criteria:

(1) Greater than or equal to 34+0 gestational weeks and less than or equal to 35+6 gestational weeks at enrolment;

Exploratory study-specific criteria:

1. Greater than or equal to 34+0 gestational weeks and less than or equal to 38+6 gestational weeks at enrolment;
2. Confirmed diagnosis of GDM or having diabetes mellitus.

Exclusion Criteria:

1. Multiple pregnancies (three or more pregnancies)
2. For subjects who are unable to be included in this study in the following cases:
3. Pregnant women with ectopic pregnancy
4. Fetal distress, severe infectious (e.g. sepsis, infectious shock) disease, fever;
5. Those who have taken glucocorticoid drugs within 2 weeks before joining the clinical trial;
6. Those who took clindamycin during the study period;
7. Those with congenital foetal anomalies or foetal hypoxia occurring in early pregnancy;
8. Patients with convulsions;
9. Those with a history of HIV/HCV/hepatitis A, substance abuse;
10. Chorioamnionitis, endometritis;
11. Placental abruption, use of surfactant, severe intrauterine haemorrhage;
12. Pregnant women with cervical dilatation greater than or equal to 4 cm or ultrasonographic neck length greater than or equal to 20 mm;
13. Pregnant women taking food or drugs during the study period that may affect foetal safety;
14. Pregnant women participating in other clinical trials.
15. Gestational diabetes mellitus and patients with diabetes mellitus (exclusion criteria for half-dose studies only).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory distress syndrome | Detection and evaluation of the newborn within 24 hours of the end of delivery
  Dependent on clinical presentation, arterial blood gas analysis, and chest X-ray. (1) progressive dyspnoea, expiratory groaning, inspiratory trigonocephaly, cyanosis, and markedly reduced or absent breath sounds on lung auscultation that appeared shortly after birth; (2) lung X-ray changes typical of RDS, with diffuse fine-grained reticulated ground-glass shadows accompanied by bronchial insufflation signs; and (3) exceptions to dyspnoea caused by simple severe pneumonia, meconium aspiration or pulmonary haemorrhage, etc.
PK parameters (analysed in conjunction with population pharmacokinetic (PPK) modelling): area under the blood concentration curve, Cmax, Tmax, Kel, t1/2, CL, VZ | 2±0.5 h, 12 h after first dose
  Blood concentrations of dexamethasone and its metabolites and foetal blood concentrations
Pharmacodynamics | In the course of pregnancy (GW8-delivery), the blood samples were collected every 2 weeks on average, and the blood samples were collected during each delivery and at the time of delivery, and the exact time of delivery was slightly adjusted according to
  Biomarker assay and measurement of placental P-gp regulatory sensitive factor pregnancy blood concentrations.
Measurability indicators | during labour
  Measurable indicators: neonatal head circumference, length, weight, blood pressure (diastolic/systolic);
Blood biochemistry findings in newborns | during labour
  Blood glucose concentration, blood triglyceride concentration, etc.
DEX potential safety marker test | during labour
  Maternal blood and umbilical vein blood were collected at the time of delivery and concentrations of potentially toxic biomarkers (e.g. ACTH, CORT, GABA, GAD67) were measured

IPD SHARING:
Plan to Share IPD: No